CLINICAL TRIAL: NCT03100227
Title: (18)F-FDG PET Database of Adult Healthy Individuals for Clinical Studies in Epileptic Patients
Brief Title: (18)F-FDG PET Database of Adult Healthy Individuals
Acronym: BDD-FDG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL16_0689
Record Dates: First submitted 2017-02-23; First posted 2017-04-04 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Healthy
MeSH Terms: interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PET [18F] FDG (Active Comparator): Each subject will have a PET scan at [18F] FDG.The raw imaging data obtained from these controls will be post-processed using the Statistical Parametric Mapping software. Schematically, the data of each control will be normalized in the same anatomical space, then smoothed and averaged between the different controls. This will make it possible to constitute the normative database.
  Interventions: Other: PET [18F] FDG; Other: Anatomical MRI
- Review test-retest (Sham Comparator): Of the 40 volunteers included, 10 will have test-retest exams (2 separate exams every 15 days).
  Interventions: Other: PET [18F] FDG; Other: Anatomical MRI

INTERVENTIONS:
Other: PET [18F] FDG — Measurement of carbohydrate metabolism at the individual level. Standardization of the individual imaging data in a standard anatomical space and then calculation of an average image through the group-level controls.
Other: Anatomical MRI — All subjects will benefit from a 3D anatomical MRI to control the normality of their MRI and an automatic segmentation of 73 brain regions by multi-atlas segmentation.

SUMMARY:
Epilepsy is the most common chronic neurological disorder in the world, affecting more than 50 million people worldwide.

Approximately 35% of patients with epilepsy are refractory to all available antiepileptic drugs. Focal Hypometabolism on interictal [18F]-FDG PET is a hallmark of the Seizure Onset Zone as well as surrounding areas. Using [18F]-FDG PET is thus particularly useful to determine the seizure onset zone of epileptic patients and thus to guide surgical treatment when antiepileptic drugs fail.

Interpretation of PET images primarily relies on standard visual analysis, but statistical analysis, with the widely used Statistical Parametric Mapping (SPM) software improves the diagnostic yield of PET. Over the past years, some authors have thus reported that the use of SPM can result in greater sensitivity and specificity of PET imaging in patients with partial epilepsy.

In order to perform statistical analysis of PET images to compare brain metabolism of epileptic patients and healthy controls, it is necessary to collect a normative database of [18F]-FDG PET images in healthy controls.

The purpose of this study is (i) collect a normative database of [18F]-FDG PET images in healthy adults controls to evaluate rigorously the diagnostic value of multimodal imaging for non-invasive localization of the EZ and (ii) to evaluate the test-retest reliability of [18F]-FDG PET scanning.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult controls
* Age 20-65 years
* Signed informed consent form.

Exclusion Criteria:

* Contraindication to the MRI
* Known neurological disease
* Adult subject to legal protection measure.
* Women of childbearing age who do not have effective contraception

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2015-09-16 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Glucose Metabolism of the whole brain estimated with [18F]-FDG PET in healthy controls. | Day 1
  40 healthy controls (age range 20-65 years) will undergo [18F]-FDG PET. The Glucose Metabolism for whole brain will be determined with [18F]-FDG PET for each subject.

SECONDARY OUTCOMES:
Test-reliability | Week 2
  For each subject, we will measure Glucose Metabolism of the whole brain estimated with [18F]-FDG PET for the first PET scan and for the second PET scan and evaluate the potential difference of Glucose Metabolism between the two scans.

CONTACTS AND LOCATIONS:
Overall Officials: Julien JUNG, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zotova D, Pinon N, Trombetta R, Bouet R, Jung J, Lartizien C. GAN-based synthetic FDG PET images from T1 brain MRI can serve to improve performance of deep unsupervised anomaly detection models. Comput Methods Programs Biomed. 2025 Jun;265:108727. doi: 10.1016/j.cmpb.2025.108727. Epub 2025 Mar 31. PMID 40187100
- [Background] Merida I, Jung J, Bouvard S, Le Bars D, Lancelot S, Lavenne F, Bouillot C, Redoute J, Hammers A, Costes N. CERMEP-IDB-MRXFDG: a database of 37 normal adult human brain [18F]FDG PET, T1 and FLAIR MRI, and CT images available for research. EJNMMI Res. 2021 Sep 16;11(1):91. doi: 10.1186/s13550-021-00830-6. PMID 34529159